CLINICAL TRIAL: NCT00772330
Title: Clinical Study of the Safety and Performance of the Miami InnFocus Drainage Implant to Relieve Glaucoma Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: InnFocus Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INN003
Record Dates: First submitted 2008-10-13; First posted 2008-10-15 (Estimated); Results first posted 2021-07-14 (Actual); Last update posted 2021-07-14 (Actual); Status verified 2021-06

CONDITIONS: Glaucoma
Keywords: MIDI Arrow; Glaucoma Drainage Device; GDD; InnFocus; Glaucoma treatment
MeSH Terms: conditions — Glaucoma | interventions — Glaucoma Drainage Implants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MIDI Arrow (Experimental): Ab externo glaucoma drainage device with no reservoir
  Interventions: Device: Glaucoma Drainage Device

INTERVENTIONS:
Device: Glaucoma Drainage Device — Insertion of MIDI Arrow subconjunctivally with a fornix-based incision after pretreatment of scleral surface with 0.4 mg/mL MMC and insertion of MIDI Arrow tube through sclera into anterior chamber of eye

SUMMARY:
Assess the safety and performance of the Miami InnFocus Drainage Implant in patients suffering from glaucoma that is inadequately controlled on tolerated medical therapy with intraocular pressure greater than or equal to 18 mm Hg and less than or equal to 40 mm Hg.

DETAILED DESCRIPTION:
Unicentric, non-randomized, single arm safety and performance study which will be conducted in accordance with the applicable parts of CFR 21 and Standard EN-ISO 14155 I & II: 2003 on clinical investigations with medical devices on human subjects and recommendations guiding physicians in biomedical research involving human subjects adopted by the 18th World Medical Assembly, Helsinki, Finland, 1964 and later revisions

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age 18 to 85 years, inclusive
* Glaucoma that is inadequately controlled on tolerated medical therapy with intraocular pressure greater than or equal to 18 mm Hg and less than or equal to 40 mm Hg.
* Patient must have signed informed consent form

Exclusion Criteria:

* Unwilling or unable to give informed consent or unable to return for scheduled protocol visits
* Pregnant or nursing women
* No light perception
* Active iris neovascularization or active proliferative retinopathy
* Iridocorneal endothelial syndrome
* Epithelial or fibrous downgrowth
* Aphakia (without pseudophakia)
* Vitreous in anterior chamber for which a vitrectomy is anticipated
* Chronic or recurrent uveitis
* Severe posterior blepharitis
* Unwilling to discontinue contact lens use after surgery
* Previous ophthalmic surgery, excluding uncomplicated phacoemulsification (cataract) surgery or corneal refractive surgery
* Need for glaucoma surgery combined with other ocular procedures other than cataract surgery (i.e., penetrating keratoplasty or retinal surgery) or anticipated need for additional ocular surgery
* Known allergy to Mitomycin C (MMC) drug.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2007-10; Primary Completion 2016-11 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Juan F Batlle, MD, Principal Investigator — Laser Center, Santo Domingo, Dominican Republic
Locations (1):
- Laser Center, Santo Domingo, Dominican Republic

REFERENCES:
- [Derived] Garcia-Feijoo J, Batlle JF, Aptel F, Lachkar Y, Riss I, Sadruddin O, Nguyen T, Beckers HJM. Pooled Analysis of Three MicroShunt Studies in Primary Open-Angle Glaucoma Evaluating Different Concentrations of Applied Mitomycin C. Ophthalmol Ther. 2025 Jul;14(7):1533-1549. doi: 10.1007/s40123-025-01149-4. Epub 2025 May 23. PMID 40408035
- [Derived] Batlle JF, Corona A, Albuquerque R. Long-term Results of the PRESERFLO MicroShunt in Patients With Primary Open-angle Glaucoma From a Single-center Nonrandomized Study. J Glaucoma. 2021 Mar 1;30(3):281-286. doi: 10.1097/IJG.0000000000001734. PMID 33137019

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This report presents data for 23 patients (Patients 13 to 35), who were implanted with the MicroShunt (one eye implanted per patient)
Groups:
- MIDI Arrow: Eligible patients with POAG were implanted with a MicroShunt in the anterior chamber of the eye
Period: Overall Study
Arm/Group | MIDI Arrow
Started | 23
Completed | 20
Not Completed | 3
Not completed — Lost to Follow-up | 3

BASELINE CHARACTERISTICS:
Population: Intention to Treat (ITT) Population: all enrolled patients.
Groups:
- Patient With Primary Open Angle Glaucoma (POAG): Patient with primary open angle glaucoma (POAG) inadequately controlled on tolerated medical therapy with IOP ≥ 18mmHg and ≤ 40 mmHg
Arm/Group | Patient With Primary Open Angle Glaucoma (POAG)
Number analyzed (Participants) | 23
Age, Continuous [Mean (Full Range); unit: years] | 59.8 [30 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 15
Region of Enrollment [Count of Participants; unit: Participants]
  Dominican Republic | 23

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Performance Success
Description: Success: IOP < 15 mmHg or IOP reduced from baseline (pre-operative level) by ≥ 20% (without glaucoma reoperation, such as a trabeculectomy to improve aqueous drainage or implantation of another drainage implant).
Time Frame: Day 1, Day 7, Week 3, Week 6, Month 3, Month 9, Month 12, Month 24, Month 36, Month 48 and Month 60
Population: Intention to Treat (ITT) Population: all enrolled patients.
Measure: Count of Participants; unit: Participants
Groups:
- To Assess Safety and Performance of the MIDI Arrow in Patients w Glaucoma: To Assess safety and performance of the MIDI arrow in patients suffering from Glaucoma inadequately controlled on medical therapy with IOP >/= 18mmHg and </= 40mmHg
Arm/Group | To Assess Safety and Performance of the MIDI Arrow in Patients w Glaucoma
Number analyzed (Participants) | 23
Participants
  Day 1 | 22
  Day 7 | 23
  Week 3 | 23
  Week 6 | 23
  Month 3 | 22
  Month 9 | 23
  Month 12 | 22
  Month 24 | 21
  Month 36 | 20
  Month 48 | 17
  Month 60 | 18

2. Secondary Outcome: Maintenance of Pressure Control
Description: Maintenance of pressure control throughout the follow-up period, as measured by IOP at each post-operative visit
Time Frame: Day 1, Day 7, Week 3, Week 6, Month 3, Month 9, Month 12, Month 24, Month 36, Month 48 and Month 60
Population: Intention to Treat (ITT) Population: all enrolled patients
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | To Assess Safety and Performance of the MIDI Arrow in Patients w Glaucoma
Number analyzed (Participants) | 23
mmHg
  Baseline IOP | 23.78 (5.342)
  Day 1 | 9.6 (5)
  Day 7 | 7.8 (2.9)
  Week 3 | 7.4 (2.26)
  Week 6: number analyzed (Participants) | 22
  Week 6 | 8.9 (3.81)
  Month 3 | 10.8 (6.07)
  Month 6 | 12 (6.17)
  Month 9 | 11.2 (3.15)
  Month 12 | 11.3 (4.07)
  Month 24: number analyzed (Participants) | 22
  Month 24 | 12 (3.64)
  Month 36: number analyzed (Participants) | 21
  Month 36 | 11.8 (6.58)
  Month 48: number analyzed (Participants) | 14
  Month 48 | 12 (3.52)
  Month 60: number analyzed (Participants) | 18
  Month 60 | 11.5 (4.89)

3. Other Pre Specified Outcome: Procedure Feasibility
Description: Defined by ease of insertion of the device into the anterior chamber, based on an Investigator evaluation rating (5-point scale, with 1 being difficult and 5 being easy);
Time Frame: Day 1
Population: Intention to Treat (ITT) Population: all enrolled patients.
Measure: Number; unit: Participants
Arm/Group | MIDI Arrow
Number analyzed (Participants) | 23
Participants
  1 - Difficult | 0
  2 | 0
  3 | 0
  4 | 6
  5 - Easy | 17

4. Other Pre Specified Outcome: Time (in Minutes) Taken for the Procedure
Description: The mean surgical procedure time from the time the incision was made in the conjunctiva to the time peritomy closure
Time Frame: Day 1
Population: Intention to Treat (ITT) Population: all enrolled patients.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | MIDI Arrow
Number analyzed (Participants) | 23
Minutes | 25.3 (7.82)

5. Other Pre Specified Outcome: Visual Acuity
Description: Visual acuity measured at each post-operative visit from baseline.
Time Frame: Day 1, Day 7, Week 3, Week 6, Month 3, Month 9, Month 12, Month 24, Month 36, Month 48 and Month 60
Population: Intention to Treat (ITT) Population: all enrolled patients.
Measure: Mean (Standard Deviation); unit: LogMar
Arm/Group | MIDI Arrow
Number analyzed (Participants) | 22
LogMar
  Baseline | .94 (1.143)
  Day 1 | 1.28 (1.203)
  Day7: number analyzed (Participants) | 20
  Day7 | .99 (1.023)
  Week 3 | .87 (.991)
  Week 6: number analyzed (Participants) | 20
  Week 6 | .76 (1.031)
  Month 3 | .92 (1.226)
  Month 6 | .85 (1.211)
  Month 9 | .85 (1.176)
  Month 12 | .79 (1.113)
  Month 24: number analyzed (Participants) | 21
  Month 24 | .90 (1.151)
  Month 36: number analyzed (Participants) | 18
  Month 36 | .69 (.992)
  Month 48: number analyzed (Participants) | 12
  Month 48 | .44 (.741)
  Month 60: number analyzed (Participants) | 14
  Month 60 | .43 (.909)

6. Other Pre Specified Outcome: Visual Field
Description: Visual field measure at each post op visit. Data not available for summary as per CSR
Time Frame: 60 Months
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Incidence of Glaucoma Re-operation
Description: Cases requiring glaucoma re-operation
Time Frame: 60 Months
Population: Intention to Treat (ITT) Population: all enrolled patients.
Measure: Number; unit: participants
Arm/Group | MIDI Arrow
Number analyzed (Participants) | 23
participants | 2

8. Other Pre Specified Outcome: Glaucoma Supplemental Medication
Description: The number of glaucoma supplemental medications required after the MicroShunt procedure.
Time Frame: Day 1 thru Month 3, Month 6, Month 9, Month 12, Month 24, Month 36, Month 48 and Month 60
Population: Intention to Treat (ITT) Population: all enrolled patients.
Measure: Median (Full Range); unit: Medications
Groups:
- The Number of Glaucoma Supplemental Medication: the number of glaucoma supplemental medications required after the MicroShunt procedure
Arm/Group | The Number of Glaucoma Supplemental Medication
Number analyzed (Participants) | 23
Medications
  Baseline | 2 [1 to 4]
  Day 1 thru Month 3 | 0 [0 to 0]
  Month 6 | 0 [0 to 2]
  Month 9 | 0 [0 to 2]
  Month 12 | 0 [0 to 3]
  Month 24: number analyzed (Participants) | 22
  Month 24 | 0 [0 to 3]
  Month 36: number analyzed (Participants) | 21
  Month 36 | 0 [0 to 4]
  Month 48: number analyzed (Participants) | 14
  Month 48 | 0 [0 to 3]
  Month 60: number analyzed (Participants) | 18
  Month 60 | 0 [0 to 4]

9. Other Pre Specified Outcome: Implant Migration
Description: Incidence of implant migration. None reported
Time Frame: 60 Months
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Implant Encapsulation
Description: Incidence of implant encapsulation. None reported
Time Frame: 60 Months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were reported up to 60 months of follow up.
Description: Any untoward medical occurrence in a subject
Arm/Group | Patient With Primary Open Angle Glaucoma (POAG)
All-Cause Mortality (participants affected / at risk) | 0/23
Serious Adverse Events (participants affected / at risk) | 8/23
Other Adverse Events (participants affected / at risk) | 21/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patient With Primary Open Angle Glaucoma (POAG) (N=23)
Posterior capsule opacification (Eye disorders) | 2 (2)
Intraocular pressure increased (Investigations) | 4 (6)
Eye operation complication (Injury, poisoning and procedural complications) | 1 (1)
Iris adhesions (Eye disorders) | 1 (1)
Tenon's cyst (Injury, poisoning and procedural complications) | 1 (1)
Cataract (Eye disorders) | 2 (2)
Malignant Glaucoma (Eye disorders) | 1 (1)
Angina (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patient With Primary Open Angle Glaucoma (POAG) (N=23)
Anterior chamber inflammation (Eye disorders) | 1 (11)
Choroidal effusion (Eye disorders) | 2 (2)
Conjunctival bleb (Eye disorders) | 2 (3)
Conjunctival hyperaemia (Eye disorders) | 1 (1)
Corneal oedema (Eye disorders) | 5 (5)
Corneal striae (Eye disorders) | 2 (2)
Dry eye (Eye disorders) | 1 (1)
Eye pain (Eye disorders) | 4 (5)
Flat anterior chamber of eye (Eye disorders) | 3 (3)
Hypotony of eye (Eye disorders) | 4 (4)
Iris adhesions (Eye disorders) | 2 (2)
Lacrimation increased (Eye disorders) | 2 (2)
Meibomianitis (Eye disorders) | 1 (1)
Posterior capsule opacification (Eye disorders) | 3 (3)
Vitreous haemorrhage (Eye disorders) | 1 (1)
Conjunctival filtering bleb leak (Injury, poisoning and procedural complications) | 1 (1)
Eye operation complication (Injury, poisoning and procedural complications) | 4 (4)
Hyphaema (Injury, poisoning and procedural complications) | 3 (3)
Ocular procedural complication (Injury, poisoning and procedural complications) | 1 (1)
Tenon's cyst (Injury, poisoning and procedural complications) | 2 (2)
Intraocular pressure increased (Investigations) | 6 (11)
Visual field defect (Nervous system disorders) | 1 (1)
Device deployment issue (Product Issues) | 3 (3)
Device occlusion (Product Issues) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes